CLINICAL TRIAL: NCT04638322
Title: Effects of a High Intensity Interval Functional Training Program on the Cognitive and Functional Capabilities of Older Adults With Mild Cognitive Impairment.
Brief Title: Effects of Functional Training by High Intensity Intervals in Older Adults With Mild Cognitive Impairment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Agustín Aibar Almazán, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: University of Jaén (2020)
Record Dates: First submitted 2020-10-27; First posted 2020-11-20 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Quality of Life; Aging

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The assignment to the groups will be of simple random type and hidden. Those responsible for admitting patients to the intervention phase will not know what group has been assigned each. This assignment will be made in advance by a researcher who will not intervene in the later stages of evaluation, intervention, data recording and elaboration of database. The assignment will be communicated through sealed and totally opaque envelopes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIFT Group (Experimental): This group receives physical training based on exercises of high intensity interval functional training.
  Interventions: Other: HIFT Group
- No intervention group (No Intervention): This group does not receive any treatment.

INTERVENTIONS:
Other: HIFT Group — An experimental group (EG) that after an initial evaluation will be subjected to a physical training program based on the HIFT method, for 12 weeks with 2 weekly sessions (Tuesday and Thursday), with a duration of 45 min per session. Once the intervention is finished, you will undergo a final evaluation to see if there is a difference or not with the results obtained at the beginning.
  Arms: HIFT Group

SUMMARY:
To analyze the effects of a high intensity interval functional training program (HIFT), in the cognitive and functional capacities of Colombian older adults with mild cognitive impairment.

DETAILED DESCRIPTION:
This is a randomized clinical trial of single-blind with 2 arms (Control group and experimental group), in which a pre-treatment-postest design has been used.

The study will define two groups:

A control group (CG) that will not be submitted to treatment, which will be evaluated in the pre and post phase of the study. Participants assigned to this group will receive general advice on the positive effects of regular physical activity and will be given a guide to recommendations for promoting physical activity.

An experimental group (GE) that after an initial evaluation will undergo a physical training program based on high intensity interval functional training exercises.

Once the intervention is finished, it will be submitted to a final evaluation to see if there is a difference or not with the results obtained at the beginning.

ELIGIBILITY:
Inclusion Criteria:

* More than 60 years
* Adults with mild cognitive impairment
* Not participating in any physical exercise program
* Sufficient physical autonomy to participate in the physical activities required by the study
* Have no signs of dementia (<26 on MoCA)
* Be able to understand instructions, programs and protocols.

Exclusion Criteria:

* Contraindications for conducting physical tests
* Diseases that limit cognitive performance and physical activity.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
MoCA (Montreal Cognitive Assessment) | Up to twelve weeks.
  Instrument that examines the skills of attention, concentration, executive functions, memory, language, visuoconstructive abilities, calculation and orientation and the maximum score is 30.
TMT (Trail Making Test) | Up to twelve weeks.
  It is used to assess executive function. It measures timed motor and visual tasks, and is divided into two tests: Part A (TMTA), which assesses speed and psychomotor attention and requires connecting consecutively numbered circles; and Part B (TMTB), which tests executive function and requires connecting alternating circles of numbers and letters. Longer completion times indicate poor performance.
Isaacs test | Up to twelve weeks.
  Instrument used to assess verbal fluency. Participants have 60 seconds to generate as many words as possible within a given semantic category (animals, colors, fruits, and cities). The maximum score is 40 points (with a maximum of 10 per category). The higher the score, the better the level of verbal fluency.Instrument used to assess verbal fluency. Participants have 60 seconds to generate as many words as possible within a given semantic category (animals, colors, fruits, and cities). The maximum score is 40 points (with a maximum of 10 per category). The higher the score, the better the level of verbal fluency.
SFT (Senior Fitness Test) | Up to twelve weeks.
  Instrument used to assess functional abilities. It consists of the following tests: muscle strength (upper and lower limbs), aerobic endurance, flexibility (upper and lower limbs) and agility, 6-minute walk test, Sit-to-foot test using a chair (measures flexibility of the lower body, Try to clasp hands behind your back, Try to get up, walk 8 feet and sit back.
The Lawton & Brody scale | Up to twelve weeks
  Evaluates independence and functionality in instrumental activities of daily life) such as shopping, cooking, cleaning, washing, finances, medication, transportation and use of the telephone; and considers instrumental disability the inability to perform one or more activities. Each area is scored according to the description that best corresponds to the subject. Therefore, each area scores a maximum of 1 point and a minimum of 0 points. The maximum dependence would be marked by obtaining 0 points, while a sum of 8 points would express total independence.
  In a conventional way, the following classification can be assumed:
  Grades A-B or 0 - 1 points = absence of disability or mild disability. Grades C-D or 2 - 3 points = moderate disability. Grades E-G or 4 - 6 points = severe disability.
The Short Form-36 Health Survey (SF-36) | Up to twelve weeks
  Used extensively for assessing health-related quality of life. The results are values between 0 and 100. Optimal health is represented by scores of 100 and very poor health would equal 0.
The Yesavage Geriatric Depression Scale | Up to twelve weeks
  Questionnaire used to screen for depression in older people. Scores from 00 to 05 indicate Normal screening, 06 to 10 Moderate Depression screening, and 11 to 15 Severe Depression screening.
Mini-Mental State Examination (MMSE) | Up to twelve weeks
  The most widely used cognitive screening test to assess suspected symptoms consistent with cognitive impairment or dementia. Written test with a maximum score of 30. The cut-off point established for the MMSE defines "normal" cognitive function is generally set at 24, lower scores indicate more serious cognitive problems.
PSQI (Pittsburgh Sleep Quality Index) | Up to twelve weeks
  A simple and valid assessment of both sleep quality and disturbance that might affect. They consist of 10 questions divided into four subscales: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep discomfort, medication use and daytime dysfunctions, adding up to a total score. The higher value represents a worse result. Higher scores indicate poorer sleep.
Tinetti scale | Up to twelve weeks
  It is used to determine early the risk of falling in an elderly person during the year following its application. The result of both sections will be added, so that a score of less than 19 points will imply a high risk of falls, a score of 19 to 24 will reflect medium risk of falls and a score of 25 to 28 will indicate low risk of falls.
Frailty phenotype | Up to twelve weeks
  Five original characteristics are evaluated: involuntary weight loss, self-reported exhaustion, slow gait speed, weakness, and low physical activity.
The 8 foot up & go test | Up to twelve weeks
  Assesses agility and dynamic balance.
KATZ INDEX | Up to twelve weeks
  Is a widely used tool to assess the level of independency in older adults. It is scored considering the items grouped to obtain degrees A, B, C, etc., of independence. It is observed that 0 points are equal to grade A, 1 point to grade B, 2 points to grade C, 3 points to grade D, and so on.
  In a conventional way, the following classification can be assumed:
  Grades A-B or 0 - 1 points = absence of disability or mild disability. Grades C-D or 2 - 3 points = moderate disability. Grades E-G or 4 - 6 points = severe disability.
Chair sit and reach test | Up to twelve weeks
  To test low back and hamstring flexibility.
Back scratch test | Up to twelve weeks
  To measure general shoulder range of motion.

SECONDARY OUTCOMES:
D2 test | Up to twelve weeks.
  Time-limited test to measure concentration. The test measures the processing speed, the following of instructions and the goodness of the execution in a task of discrimination of similar visual stimuli and that, therefore, allow the estimation of attention and concentration.
DSST (The Digit Symbol Substitution Test) | Up to twelve weeks.
  Cognitive test to assess processing speed presented on a single sheet of paper that requires a subject to match symbols with numbers according to a key located at the top of the page. The subject copies the symbol into spaces below a row of numbers. The number of correct symbols within the allowed time, usually 90-120 seconds, constitutes the score.
Mindful Attention Awareness Scale (MAAS) | Up to twelve weeks.
  It evaluates, in a global way, the dispositional capacity of an individual to be attentive and aware of the experience of the present moment in everyday life. The scale is a 15-item univariate self-report with a view of the mindfulness construct centered on the attention / consciousness variable.
Handgrip Strength | Up to twelve weeks.
  Dynamometer will be employed to assess hand grip stregth.
BMI (Body Mass Index) | Up to twelve weeks.
  Is calculated from the formula, Weight (kg) / Height2 (m2), whose unit is kg/m2. It is a rough indicator of total body fat
Waist circumference | Up to twelve weeks.
  Is used to assess central fat distribution and degree of abdominal obesity
Waist-to-hip ratio | Up to twelve weeks.
  Is the dimensionless ratio of the circumference of the waist to that of the hips. This is calculated as waist measurement divided by hip measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Casa de los Tiempos, Cali, Valle del Cauca Department, Colombia